CLINICAL TRIAL: NCT00731172
Title: A Pilot Single Center,Randomized,Double Blind Placebo Controlled Study to Assess the Safety,Tolerability and Efficacy of Copaxone in Inducing Remission in Patients With Moderately Active Crohn's Disease.
Brief Title: A Double Blind Placebo Control Study to Assess the Safety,Tolerability and Efficacy of Copaxone in Crohn's Disease
Acronym: Cop1CD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry); Medtronic - MITG (Industry)
Responsible Party: Iris Dotan, MD, Tel Aviv sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-ID-037-CTIL
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Crohns Disease
Keywords: crohns disease
MeSH Terms: conditions — Crohn Disease | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 20 mg copaxone(glatiramer acetate)subcutaneous injection(daily through week 12)
  Interventions: Drug: glatiramer acetate
- 2 (Placebo Comparator): placebo subcutaneous injection(daily through week 12)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glatiramer acetate — 20 mg daily subcutaneous injection through week 12
  Arms: 1
Drug: placebo — subcutaneous daiky injection through week 12
  Arms: 2

SUMMARY:
phase 2 study. Target disease: Crohn's disease.

Rational and relevance to IBD patients:

Copaxone is known for its high safety profile and for acting as an effective immunomodulatory agent for the treatment of MS. . In experimental models of IBD, a beneficial effect of Copaxone was demonstrated where significant amelioration of macroscopic colonic damage, preservation of the microscopic colonic structure, reduced weight loss, and improved long-term survival in treated compared with untreated mice was demonstrated. In addition, Copaxone suppressed the proliferation of local mesenteric lymphocytes to syngeneic colon extract, significantly reduced the overall secretion of TNF-α and induced the secretion of transforming growth factor (TGF)-β. The ability of Copaxone to effectively modulate the clinical manifestations and the detrimental immune response involved in experimental colitis, together with its high safety profile support its potential effect as a new treatment for CD.

Patients: patients with moderately active Crohn's disease as indicated by a CDAI 220 - 450, whose diagnosis was done more than 3 months before enrollment.

Study objectives: to test the efficacy and safety of Copaxone in CD patients.

Study design: This will be a single center, randomized, double blind placebo controlled phase 2 study.

Subjects will be assessed for study eligibility 1 to 2 weeks prior to baseline Eligible patients will be enrolled into the study after signing an informed consent form and allocated in a 1.5:1 ratio to receive either Copaxone or placebo. A total of 50 patients will be recruited.

Subcutaneous injections (Copaxone or Placebo) will be administered daily through week 12. Patient assessment of safety and efficacy will be made at weeks 0,4,8,12 and 16.

At week 12 non-responders would be offered an open label arm with daily Copaxone 20mg for the next 12 weeks

DETAILED DESCRIPTION:
Data evaluation: Evidence of therapeutic benefit and safety will be evaluated by the following assessments:

Clinical assessments:

* Crohn's disease activity will be assessed by components of the CDAI.
* Mucosal healing will be assessed by VCE (data will be quantitated using the Lewis score). Patients requiring colonoscopy according to Physicians decision would also be offered to participate in an endoscopic mucosal healing evaluation substudy. Patients participating will undergo colonoscopy and biopsies at the beginning (screening±1 week) and the end (week 12±1 week) of the treatment period. Endoscopic damage will be assessed using the CDEIS
* Mean (median) doses of corticosteroids and the average total aggregate dose of corticosteroids received per patient during the trial will be assessed.
* Quality of life will be assessed by components of the Inflammatory Bowel Disease Questionnaire(IBDQ).

Safety:

* AE incidence
* Physical examination
* Clinical laboratory values
* Vital signs

Tolerability and Safety:

* Adverse events, dropout rate will be registered.
* Proportion of subjects who prematurely discontinue the study.
* Proportion of subjects who prematurely discontinue the study due to Aes
* Time to premature discontinuation
* Time to premature discontinuation due to Aes.

Immunologic assessment (including lymphocyte proliferation and cytokine secretion assays) will be performed at the baseline visit as well as weeks 4 and 12 and 16. Serum samples for cytokine studies 24 hours after first injection would also be collected.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the trial, patients must meet all of the following criteria;

1. Are 18-70 years old at the time of screening; may be male or female.
2. Have Crohn's disease, diagnosed more than 3 months before enrollment and confirmed by endoscopy, radiology or surgery. Documentation should be performed within 36 months prior to screening.
3. Moderately active Crohn's disease as indicated by a CDAI 220 - 450.
4. Are able to adhere to the following concomitant medication requirements:

   1. Patients must never have received treatment with Copaxone.
   2. Patients taking 5-ASA compounds must have been taking the drug for at least 4 weeks with a stable dosage for at least 2 weeks prior to screening.
   3. Patients taking oral corticosteroids must have been taking the drug for at least 4 weeks prior to screening. These patients must be with a stable dose of up to20 mg prednisone/day or equivalent, or up to 6 mg budesonide/day for at least 2 weeks prior to screening.

      Inhaled or topical steroids are allowed.
   4. Patients taking AZA or 6MP must be on a stable dose for at least 12 weeks prior to screening.
   5. Patients taking antibiotic therapy for CD must be on a stable dose for at least 2 weeks prior to screening.
5. Negative stool cultures for enteric pathogens (Salmonella, Shigella, Campylobacter) and negative Clostridium difficile toxin assay in stool.
6. Women and men of childbearing potential must use medically acceptable methods of contraception [surgical sterilization, IUD, hormonal preparations, or double barrier method (e.g. condom or diaphragm, and spermicide)] throughout the study.
7. Patients are able to self-inject or have a designee or healthcare professional who can inject the study medication daily.
8. Patients are willing and able to provide written informed consent.

Exclusion Criteria:

1. Diagnosis of indeterminate, microscopic, lymphocytic, collagenous, or ulcerative colitis.
2. Subjects with clinically significant active systemic infection.
3. Subjects who in the opinion of the investigator have another clinically significant or unstable medical or surgical condition such as: cardiovascular, pulmonary, hepatic, renal, autoimmune, endocrine, metabolic or malignancy or any other condition that places the subject at undue risk by participating in the study.
4. Short bowel syndrome or a bowel surgery within 3 month before randomization.
5. Clinically significant obstructive symptoms with radiologic evidence of intestinal strictures. Ileostomy, colostomy, or parenteral nutrition Subjects who have fistula with abscess formation.
6. The use of the following medications within the last 12 weeks prior to screening: TNF-a antibodies, Thalidomide, Methotrexate, Cyclosporine, Tacrolimus, or Mycophenolate Mofetil.
7. The use of more than 100mg/d Aspirin.
8. Use of another investigational drug within 3 months before screening.
9. Pregnant or lactating woman.
10. Concomitant substance or alcohol abuse.
11. Subjects with known sensitivity to mannitol.
12. Subjects unable to self-inject or do not have a designee or healthcare professional who can inject the study medication.
13. Subject unable to comply with the planned schedule of study visits and study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints: The proportion of patients at clinical remission (CDAI<150) | week 12.

SECONDARY OUTCOMES:
Proportion of patients at clinical remission | at weeks 4 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Weizmann Institute of Science, Rehovot
  - Tel Aviv Sourasky medical center, Tel Aviv

REFERENCES:
- [Background] Aharoni R, Kayhan B, Arnon R. Therapeutic effect of the immunomodulator glatiramer acetate on trinitrobenzene sulfonic acid-induced experimental colitis. Inflamm Bowel Dis. 2005 Feb;11(2):106-15. doi: 10.1097/00054725-200502000-00003. PMID 15677903
- [Background] Aharoni R, Kayhan B, Brenner O, Domev H, Labunskay G, Arnon R. Immunomodulatory therapeutic effect of glatiramer acetate on several murine models of inflammatory bowel disease. J Pharmacol Exp Ther. 2006 Jul;318(1):68-78. doi: 10.1124/jpet.106.103192. Epub 2006 Apr 19. PMID 16624971